CLINICAL TRIAL: NCT03547401
Title: Ankle/Brachial Non-Invasive Blood Pressure Difference During General Anesthesia: a Prospective Cohort Observational Study in Young Healthy Patients
Brief Title: Ankle/Brachial Non-Invasive Blood Pressure Difference During General Anesthesia
Status: Completed | Type: Observational
Sponsor: Philippe VAN DER LINDEN (Other)
Responsible Party: Sponsor-Investigator, Philippe VAN DER LINDEN, Professor, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-ABI
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia: Patient (15 to 40 years old) undergoing elective surgery requiring general anesthesia in supine position.
  Interventions: Device: Ankle Non-invasive Blood pressure measurement; Device: Arm Non-invasive Blood pressure measurement

INTERVENTIONS:
Device: Ankle Non-invasive Blood pressure measurement — Non-invasive blood pressure measured simultaneously at the arm (model IntelliVue M8105a MP5 Phillips, calibrated).
Device: Arm Non-invasive Blood pressure measurement — Non-invasive blood pressure measured simultaneously at the ankle (model IntelliVue M8105a MP5 Phillips, calibrated).

SUMMARY:
Brachial non-invasive blood pressure (NIBP) monitoring is recommended as part of the American Society of Anesthesiology (ASA) basic monitoring package. Although brachial NIBP is often practical, some surgeries and patients may require NIBP measurement elsewhere (e.g. the ankle).

Several studies have shown that ankle NIBP overestimates brachial NIBP measurements. Algorithms have been proposed, based on correlation studies, to estimate brachial NIBP from ankle NIBP during general anesthesia and mechanical ventilation. These algorithms, however, are based on both heterogeneous populations and surgeries.

Our aim was to determine if ankle brachial NIBP difference occurs in in young ASA physical status 1 patients undergoing general anesthesia in the supine position. We also aim to determine if this difference is constant during anesthesia or if it varies according to different predefined time points.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) pysical status score 1
* Patient undergoing elective surgery requiring general anesthesia in supine position

Exclusion Criteria:

* Patient refusal
* systemic pathology
* Body mass index (BMI) superior to 30
* Surgeon requiring a position other than supine

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient undergoing elective surgery requiring general anesthesia in supine position. American Society of Anesthesiology (ASA) pysical status score 1.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Ankle Brachial non-invasive blood pressure difference - time point 1 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, before induction of anesthesia
Ankle Brachial non-invasive blood pressure difference - time point 2 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, after induction of anesthesia
Ankle Brachial non-invasive blood pressure difference - time point 3 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, after securing airway
Ankle Brachial non-invasive blood pressure difference - time point 4 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, at surgical incision
Ankle Brachial non-invasive blood pressure difference - time point 5 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, 10 minutes after surgical incision
Ankle Brachial non-invasive blood pressure difference - time point 6 | 1 day
  Difference between the non-invasive blood pressure measured at the ankle and at the arm, at reversal of anesthesia

SECONDARY OUTCOMES:
Pain at the arm (yes/no) | 1 day
  Answer 'yes' or 'no' to the question 'pain at the arm' in postoperative period
Pain at the ankle (yes/no) | 1 day
  Answer 'yes' or 'no' to the question 'pain at the ankle' in postoperative period
Ankle Brachial NIBP difference variation | 1 day
  Determine if Ankle Brachial NIBP difference remains constant or varies during different intraoperative periods

CONTACTS AND LOCATIONS:
Overall Officials: Sean Coeckelenbergh, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkes JM, DiPalma JA. Brachial blood pressure monitoring versus ankle monitoring during colonoscopy. South Med J. 2004 Oct;97(10):939-41. doi: 10.1097/01.SMJ.0000129929.28792.77. PMID 15558917
- [Background] Drake MJ, Hill JS. Observational study comparing non-invasive blood pressure measurement at the arm and ankle during caesarean section. Anaesthesia. 2013 May;68(5):461-6. doi: 10.1111/anae.12194. Epub 2013 Mar 11. PMID 23480469
- [Background] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553